CLINICAL TRIAL: NCT05558293
Title: Impact of Periodontal Bacteria on the Effectiveness of Periodontal Therapy Outcomes in Patients With Periodontitis: A Prospective Clinical and Microbial Study
Brief Title: Impact of Periodontal Bacteria on the Effectiveness of Periodontal Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Researcher, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-2018-10
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Periodontitis
Keywords: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Intervention Model Description: Patients undergo non-surgical quadrant scaling and root planing
Who Masked: Participant, Investigator
Masking Description: Both participants and clinicians were blinded to group and treatment assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periodontitis quadrant Scaling root planing (Placebo Comparator): Patients undergo non surgical quadrant scaling and root planing performed per quadrant
  Interventions: Procedure: Scaling and root planing
- Periodontitis full mouth scaling root planing (Active Comparator): Patients undergo non surgical full mouth scaling and root planing
  Interventions: Procedure: Scaling and root planing

INTERVENTIONS:
Procedure: Scaling and root planing — Full mouth or quadrant SRP

SUMMARY:
In light of the controversy that are already approved but that however still exists regarding the efficacy and influence of the protocols for the management of periodontitis, the aim of this study was to evaluate, at 6 months follow-up, the post-treatment clinical parameters and immunological and gingival microbial profiles in patients with periodontitis, treated by either SRP in addition to full mouth periodontal debridement.

DETAILED DESCRIPTION:
This trial was conducted in accordance with the World Medical Association's Declaration of Helsinki of 1975, and reviewed in 2008. Patients were enrolled from January 2020 to December 2022. The local ethical committee of approved the study protocol (125/PO) and each patient was carefully informed about the possible inherent risks of the study and provided their informed written consent 88 patients, aged 27 to 65 (mean age 57) were assessed for eligibility. In all subjects, subgingival plaque will acquired from 4 separate proximal periodontal sites.

ELIGIBILITY:
Inclusion Criteria:

1. good condition of general health,
2. a minimum of 2 teeth for each quadrant with a Pocket Depth (PD) ranging from 4-6 mm,
3. no involvement of the furcation,
4. a minimum of a six teeth per quadrant, respectively.

Exclusion Criteria:

1. periodontal therapy during the last 12 months,
2. assumption of antibiotics during the last 6 months,
3. pregnancy,
4. any systemic condition which might affect the effects of the study treatment,
5. previous or current radiation or immunosuppressive therapies,
6. use of mouthwash containing antimicrobials during the previous 3 months,
7. no use of hormonal contraceptives,
8. medication by anti-inflammatory and immunosuppressive drugs,
9. previous history of hard-drinking,
10. smoking,
11. class II and III tooth mobility.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Probing depth changes | 6 months
  Measurment of Probing Depth changes in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Isola, Principal Investigator — University of Catania
Locations (1):
- University of Catania, Catania, CT, Italy

IPD SHARING:
Plan to Share IPD: Yes
Sharing inflammatory results
Supporting Information: Study Protocol
Time Frame: 6 months
Access Criteria: University website and pubmed